CLINICAL TRIAL: NCT05848414
Title: Short Term Outcomes in Hospitalized Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Hassan Mohamed kotbey, Doctor, Assiut University
Other Study IDs: Liver cirrhosis mortality
Record Dates: First submitted 2023-03-28; First posted 2023-05-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-07

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be conducted to assess the baseline characteristics and evaluate the 90-day mortality of patients admitted with liver cirrhosis. Also, the study will be done to identify the risk factors of 90-day mortality.

DETAILED DESCRIPTION:
Liver cirrhosis is the end spectrum of all chronic liver diseases characterized by advanced fibrosis, scarring, and formation of regenerative nodules leading to hepatic architectural distortion.

Liver cirrhosis is a major cause of health burden worldwide. According to the Global Burden of Disease study, liver cirrhosis caused 1.2% of global disability-adjusted life years and 2% of all deaths worldwide in 2010, the 14th leading cause of mortality.

The progress rate of compensated cirrhosis to decompensated cirrhosis is approximately 58% and once it progresses to decompensated cirrhosis, its mortality rate within 5 years becomes 85% without liver transplantation. Since the progression of cirrhosis is accelerated each time a complication recurs, the management and treatment of the complication are critical in enhancing the quality of life and the life expectancy of patients .

Post-discharge outcomes are an integral component of healthcare, as they may aid in determining the success and longevity of treatment and how clinicians approach future cases .

This study will focus on the short-term outcomes of patients hospitalized with liver cirrhosis to provide insight into methods for future healthcare interventions.

ELIGIBILITY:
Inclusion Criteria:

- diagnosis of liver cirrhosis, adult (age ≥ 18 years old) and patients willing to give consent during the selected period.

Exclusion Criteria:

- Patients with ages < 18 years or patients that will be lost on follow-up will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All liver cirrhosis patients admitted to hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
evaluate the 90-day mortality of patients admitted with liver cirrhosis | 90 days
  Mortality

SECONDARY OUTCOMES:
identify the risk factors of 90-day mortalit | 90 days
  Risk factors for mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ahlam M Farghaly, Study Director — AhlamGastro2000@yahoo.com
Locations (1):
- Esraa Hassan Mohamed Kotbey, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsochatzis EA, Bosch J, Burroughs AK. Liver cirrhosis. Lancet. 2014 May 17;383(9930):1749-61. doi: 10.1016/S0140-6736(14)60121-5. Epub 2014 Jan 28. PMID 24480518